CLINICAL TRIAL: NCT05857800
Title: Exploring the Neo-Adjuvant Therapy Effects on Lung Cancer Through Monitoring and Assessment of Tumor Environment (NAT-LungMate)
Brief Title: Exploring the Neo-Adjuvant Therapy Effects on Lung Cancer Through Monitoring and Assessment of Tumor Environment
Acronym: NAT-LungMate
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: NAT-LungMate
Record Dates: First submitted 2023-04-28; First posted 2023-05-15 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer patients: Patients in LungMate clinical trial series.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Analysis of dynamic changes of lung cancer microenvironment in neoadjuvant therapy using bio-omics information collected in clinical trials.

SUMMARY:
This translational study aims to investigate how neoadjuvant therapy affects lung cancer patients by monitoring dynamic changes in the tumor environment. The study focuses on patients with histologically confirmed lung cancer, including non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC), who are eligible for neoadjuvant therapy in the LungMate clinical trial series. By analyzing intra-tumour genetic and functional heterogeneity following neoadjuvant therapy through multi-omic analysis (including genomics, transcriptomics, metabolomics and proteomics), this study could potentially identify new biomarkers or therapeutic targets that could improve lung cancer patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in LungMate clinical trial series, including:

  1. LungMate-001: Clinical study for neoadjuvant anti-PD-1 inhibitor, sintilimab, chemotherapy combined with surgery in treating phase IB - IIIA non-small cell lung cancer
  2. LungMate-002: Clinical study for neoadjuvant therapy of anti-PD-1 drug combined with radical surgery in treating phase IIb - III non-small cell lung cancer patients
  3. LungMate-003: Neoadjuvant PD-1 Antibody Plus Apatinib or Chemotherapy for Non-small Cell Lung Cancer
  4. LungMate-004: Neoadjuvant Afatinib Therapy for Potentially Resectable Stage III EGFR Mutation-Positive Lung Adenocarcinoma
  5. LungMate-005: Clinical Study of PD-L1 Antibody (TQB2450) Plus Chemotherapy (Cisplatin and Etoposide) for Previously Untreated Small Cell Lung Cancer
  6. LungMate-006: Clinical Study of PD-1 Antibody (BGB-A317) Plus Chemotherapy (Cisplatin and Etoposide) for Limited Stage Small Cell Lung Cancer
  7. LungMate-007: Neoadjuvant HS-10296 (Almonertinib) Therapy for Potential Resectable Stage III EGFR Mutation-Positive Lung Adenocarcinoma
  8. LungMate-009: Neoadjuvant Immunotherapy for Stage III Non-small Cell Lung Cancer
  9. LungMate-012: Neoadjuvant Furmonertinib Plus Bevacizumab or Furmonertinib Monotherapy for Resectable and Potentially Resectable Stage III-IVA EGFR Mutation-Positive Lung Adenocarcinoma
  10. LungMate-013: Induction Therapy With PD-1 Antibody Combined With Platinum-based Doublet Chemotherapy for Locally-advanced Non-small Cell Lung Cancer;
  11. LungMate-015: The Efficiency of Surgery and Radiotherapy After SHR-1316 (Adebrelimab) and Platinum-containing Doublet Induction Therapy for Limited-stage Small Cell Lung Cancer;
  12. Patients enrolled in the LungMate series of neoadjuvant therapy lung cancer clinical trials in the future;
* Age 18- years or older;
* Histopathologically confirmed with NSCLC or SCLC;
* Written Informed consent

Exclusion Criteria:

* The patients who failed to meet clinical trial screening criteria and those who dropped out of the clinical trial;
* Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
* The patient suffered from other cancers besides NSCLC (except cervical carcinoma in situ, cured basal cell carcinoma, and bladder epithelial tumor [including Ta and Tis]) within 5 years before the trial;
* The patient is a carrier of active hepatitis B, hepatitis C or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer who received neoadjuvant therapy and enrolled in the LungMate clinical trial series.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2033-05-25 (Estimated); Study Completion 2033-05-25 (Estimated)

PRIMARY OUTCOMES:
Intratumour heterogeneity index | From trial activation until trial closure (approximately 15 May 2033)
  To validate ITH index as an independent biomarker of response to neoadjuvant therapy in patients with lung cancer mutation in a gene of interest through multi-omic analysis (genomics, transcriptomics, metabolomics, proteomics) based on sequential sampling over time.
  Outcomes will be quantified using descriptive statistics with the intention of providing hypothesis-generating data for use in future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Patients are given a unique identifier as soon as they are consented. All samples and data is anonymised and can only be accessed by the research team.